CLINICAL TRIAL: NCT03963063
Title: Efficacy of Perioperative Goal-directed Fluid Therapy in Preventing Cerebral Desaturation and Postoperative Cognitive Dysfunction After Beach Chair Position Shoulder Surgery
Brief Title: Neurological Effects of Goal-directed Fluid Therapy in Beach Chair Position Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 201903017RINB
Record Dates: First submitted 2019-05-21; First posted 2019-05-24 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2020-10

CONDITIONS: Postoperative Cognitive Dysfunction; Anesthesia
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non Goal-directed Care Group (Active Comparator)
  Interventions: Procedure: Non goal-directed fluid therapy
- Goal-directed Care Group (Experimental)
  Interventions: Procedure: Goal-directed fluid therapy

INTERVENTIONS:
Procedure: Goal-directed fluid therapy — Patients in the group will follow our mini-fluid challenge test goal-directed therapy protocol, maintaining:
  * individualized optimised stroke volume by mini-fluid challenge first
  * keep mean arterial pressure ≧65 mmHg
  * keep systolic blood pressure ≦140 mmHg
  * keep cardiac index ≧ 2.5 L/min/cm2
  Arms: Goal-directed Care Group
Procedure: Non goal-directed fluid therapy — Patients in the group will receive standard perioperative care at the discretion of care-giving anesthesiologist, maintaining:
  * keep mean arterial pressure ≧65 mmHg
  * keep systolic blood pressure ≦140 mmHg
  Arms: Non Goal-directed Care Group

SUMMARY:
Patients receiving beach chair position shoulder surgery are vulnerable to perioperative cerebral desaturation, which is reported to be a risk factor for postoperative cognitive dysfunction. Investigators design this study to test the efficacy of perioperative goal-directed therapy in preventing cerebral desaturation and postoperative cognitive dysfunction in patients receiving beach chair position shoulder surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving scheduled beach chair position shoulder surgery

Exclusion Criteria:

* pregnant women
* patients in intensive care units
* patients with respiratory failure [forced expiratory volume at one second (FEV1)/ forced vital capacity (FVC) < 70 % and FEV1 < 50%]
* patients with heart failure(NYHA score =III、IV)
* patients with chronic kidney disease (eGFR< 60 ml.min-1.1.73m-2)
* patients with liver failure
* patients with ongoing infection
* patients allergic to voluven

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
duration of cerebral desaturation events | 3 hours
  patients will be monitored with bilateral cerebral oxymetry, and investigators will compare the duration of cerebral desaturation events

SECONDARY OUTCOMES:
incidence of cerebral desaturation events | 3 hours
  patients will be monitored with bilateral cerebral oxymetry, and investigators will compare the incidence of cerebral desaturation events
postoperative cognitive dysfunction assessed by the Taiwan version of questionnaire Qmci | 3 days
  Qmci is a screening assessment developed to detect mild cognitive impairment. It's a 100-point test administered in approximately 10 minutes. A score of 60 or over is considered to be normal. The validity of the Taiwan version of Qmci has been established.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Yu Wu, Ph.D., Study Director — National Taiwan University Hospital
Locations (1):
- Department of Anesthesiology, National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alam A, Hana Z, Jin Z, Suen KC, Ma D. Surgery, neuroinflammation and cognitive impairment. EBioMedicine. 2018 Nov;37:547-556. doi: 10.1016/j.ebiom.2018.10.021. Epub 2018 Oct 19. PMID 30348620
- [Background] Rappold T, Laflam A, Hori D, Brown C, Brandt J, Mintz CD, Sieber F, Gottschalk A, Yenokyan G, Everett A, Hogue CW. Evidence of an association between brain cellular injury and cognitive decline after non-cardiac surgery. Br J Anaesth. 2016 Jan;116(1):83-9. doi: 10.1093/bja/aev415. PMID 26675953
- [Result] Meex I, Vundelinckx J, Buyse K, Deburggraeve F, De Naeyer S, Desloovere V, Anne L, Truijen J, Vander Laenen M, Heylen R, De Deyne C, Jans F. Cerebral tissue oxygen saturation values in volunteers and patients in the lateral decubitus and beach chair positions: a prospective observational study. Can J Anaesth. 2016 May;63(5):537-43. doi: 10.1007/s12630-016-0604-3. Epub 2016 Feb 4. PMID 26846619
- [Result] Aguirre J, Borgeat A, Trachsel T, Cobo Del Prado I, De Andres J, Buhler P. Cerebral oxygenation in patients undergoing shoulder surgery in beach chair position: comparing general to regional anesthesia and the impact on neurobehavioral outcome. Rev Esp Anestesiol Reanim. 2014 Feb;61(2):64-72. doi: 10.1016/j.redar.2013.08.002. Epub 2013 Oct 9. PMID 24119783
- [Result] Aguirre JA, Etzensperger F, Brada M, Guzzella S, Saporito A, Blumenthal S, Buhler P, Borgeat A. The beach chair position for shoulder surgery in intravenous general anesthesia and controlled hypotension: Impact on cerebral oxygenation, cerebral blood flow and neurobehavioral outcome. J Clin Anesth. 2019 Mar;53:40-48. doi: 10.1016/j.jclinane.2018.09.035. Epub 2018 Oct 4. PMID 30292739
- [Result] Ni C, Xu T, Li N, Tian Y, Han Y, Xue Q, Li M, Guo X. Cerebral oxygen saturation after multiple perioperative influential factors predicts the occurrence of postoperative cognitive dysfunction. BMC Anesthesiol. 2015 Oct 26;15:156. doi: 10.1186/s12871-015-0117-6. PMID 26503361
- [Result] Zhang N, Liang M, Zhang DD, Xiao YR, Li YZ, Gao YG, Cai HD, Lin XZ, Lin CZ, Zeng K, Wu XD. Effect of goal-directed fluid therapy on early cognitive function in elderly patients with spinal stenosis: A Case-Control Study. Int J Surg. 2018 Jun;54(Pt A):201-205. doi: 10.1016/j.ijsu.2018.04.007. Epub 2018 Apr 17. PMID 29678619
- [Derived] Lee CT, Lin CP, Chan KC, Wu YL, Teng HC, Wu CY. Effects of Goal-Directed Hemodynamic Therapy Using a Noninvasive Finger-Cuff Monitoring Device on Intraoperative Cerebral Oxygenation and Early Delayed Neurocognitive Recovery in Patients Undergoing Beach Chair Position Shoulder Surgery: A Randomized Controlled Trial. Anesth Analg. 2023 Feb 1;136(2):355-364. doi: 10.1213/ANE.0000000000006200. Epub 2022 Sep 22. PMID 36135341